CLINICAL TRIAL: NCT03013296
Title: Delinieation of GIP's Effects During a Meal in Humans Using GIP Receptor Antagonisation (GA-4)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Lærke Smidt Gasbjerg, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UHG-CFD-GIPANTA-4
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Glucose Metabolism Disorders
Keywords: GIP; GIP receptor antagonist
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — exendin (9-39)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Saline
  Interventions: Other: Placebo
- GIP-A (Other): Infusion of GIP-A alone as study tool.
  Interventions: Other: GIP-A
- GLP-1 receptor antagonist Exendin[9-39] (Other): Infusion of GLP-1 receptor antagonist Exendin[9-39] alone as study tool.
  Interventions: Other: GLP-1 receptor antagonist Exendin[9-39]
- GIP-A + Exendin[9-39] (Other): Infusion of GIP-A + GLP-1 receptor antagonist Exendin[9-39] together as study tools.
  Interventions: Other: GIP-A + Exendin[9-39]

INTERVENTIONS:
Other: GIP-A — GIP-A
  Arms: GIP-A
Other: Placebo — Placebo
  Arms: Placebo
Other: GLP-1 receptor antagonist Exendin[9-39] — Exendin[9-39]
  Other Names: Ex(9-39)
  Arms: GLP-1 receptor antagonist Exendin[9-39]
Other: GIP-A + Exendin[9-39] — GIP-A + Exendin[9-39]
  Arms: GIP-A + Exendin[9-39]

SUMMARY:
Delinieation of GIP's effects during a meal in humans using GIP receptor antagonisation.

DETAILED DESCRIPTION:
Aim: To evaluate the role of GIPR signalling in postprandial physiology, including lipid, bone and glucose homeostasis, using a naturally occurring GIP fragment, which antagonises the GIPR.

Twelve healthy men (age 18-70 years, BMI 19-27 kg/m2) with normal kidney and liver parameters and haemoglobin levels and no first-degree relatives with type 2 diabetes will be included in a randomised, double-blinded, placebo-controlled cross-over study. Study consists of four study days with concomitant infusions of A) GIP-A, B) GLP-1 receptor antagonist Exendin[9-39], C) GIP-A + Exendin[9-39], or D) saline (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Normal kidney function, liver function and hemoglobin levels.

Exclusion Criteria:

* Medication, Diabetes type 1 or 2, BMI > 27, first degree relatives with Type 2 Diabetes

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10; Primary Completion 2017-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
C-peptide levels | 180 minutes
  Serum C-peptide AUC. Primary outcome changed during the inclusion period (original = insulin levels) due to risk of misinterpretation/diverse hepatic insulin extraction).

CONTACTS AND LOCATIONS:
Overall Officials: Fip K Knop, MD, PhD, Study Director — UHGentofte, Center for Diabetes Research
Locations (1):
- Center for Diabetes Research, Copenhagen, Gentofte, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Helsted MM, Gasbjerg LS, Lanng AR, Bergmann NC, Stensen S, Hartmann B, Christensen MB, Holst JJ, Vilsboll T, Rosenkilde MM, Knop FK. The role of endogenous GIP and GLP-1 in postprandial bone homeostasis. Bone. 2020 Nov;140:115553. doi: 10.1016/j.bone.2020.115553. Epub 2020 Jul 27. PMID 32730920
- [Derived] Gasbjerg LS, Helsted MM, Hartmann B, Sparre-Ulrich AH, Veedfald S, Stensen S, Lanng AR, Bergmann NC, Christensen MB, Vilsboll T, Holst JJ, Rosenkilde MM, Knop FK. GIP and GLP-1 Receptor Antagonism During a Meal in Healthy Individuals. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgz175. doi: 10.1210/clinem/dgz175. PMID 32077470